CLINICAL TRIAL: NCT00004984
Title: The Diabetes Prevention Trial of Type 1 Diabetes (DPT-1)
Acronym: DPT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DPT-1; U01DK060782 (NIH); U01DK060916 (NIH); U01DK060987 (NIH); U01DK061010 (NIH); U01DK061029 (NIH); U01DK061030 (NIH); U01DK061034 (NIH); U01DK061035 (NIH); U01DK061036 (NIH); U01DK061037 (NIH); U01DK061038 (NIH); U01DK061040 (NIH); U01DK061041 (NIH); U01DK061042 (NIH); U01DK061058 (NIH); U01DK061055 (NIH)
Record Dates: First submitted 2000-03-13; First posted 2000-03-14 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; insulin; prediction; prevention; C-peptide levels; insulin autoantibodies; pancreatic beta cell autoantibodies; cellular immune responses; prediction of type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The oral insulin study was masked, but the parenteral insulin study was not masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Parenteral Insulin (Experimental): High risk participants randomized to intervention
  Interventions: Drug: Parenteral Insulin
- Close Observation (Active Comparator): High risk participants randomized to observation
  Interventions: Other: Close Observation
- Oral Insulin (Experimental): Intermediate risk participants randomized to intervention
  Interventions: Drug: Oral Insulin
- Placebo (Placebo Comparator): Intermediate risk participants randomized to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Parenteral Insulin — Subcutaneous injections of recombinant human ultralente insulin in the morning and in the evening; the initial dose for each injection was 0.125 U per kilogram of body weight.
  Arms: Parenteral Insulin
Other: Close Observation — Study visits every 6 months including an oral glucose tolerance test
  Arms: Close Observation
Drug: Oral Insulin — Capsules oral insulin, 7.5 mg of recombinant human insulin crystals
  Arms: Oral Insulin
Drug: Placebo — Placebo for oral insulin
  Arms: Placebo

SUMMARY:
The Diabetes Prevention Trial of Type 1 (DPT-1) was a multicenter randomized, controlled clinical trial designed to determine whether it is possible to delay or prevent the clinical onset of type 1 diabetes through daily doses of insulin in individuals determined to be at risk for the disease. Subjects were recruited from study clinics and through media campaigns.First-degree relatives, 3 to 45 years of age, and second-degree relatives, 3 to 20 years of age, of patients with diabetes were screened for islet-cell antibodies. Those individuals found to be at high risk of diabetes were randomized to receive either close observation or low-dose parenteral insulin. Those individuals found to be at intermediate risk of diabetes are randomized to receive insulin orally or to receive placebo. Patients were followed for up to six years.

DETAILED DESCRIPTION:
The study was divided into three parts: screening, staging, and intervention. Subjects were recruited from study clinics and through media campaigns.First-degree relatives, 3 to 45 years of age, and second-degree relatives, 3 to 20 years of age, of patients with diabetes were screened for islet-cell antibodies. Those with an islet-cell antibody titer of 10 Juvenile Diabetes Foundation (JDF) units or higher were offered staging evaluations.

Staging confirmed the presence of islet-cell antibodies, measured insulin antibodies, assessed the first-phase insulin response to intravenous glucose, assessed oral glucose tolerance, and determined the presence or absence of HLA-DQA1*0102, DQB1*0602, a protective haplotype, the presence of which excluded subjects from further participation.

Islet-cell antibody-positive subjects were then defined as having a high risk of diabetes (a five-year risk of more than 50 percent) and were deemed eligible for the parenteral insulin trial if they had a first-phase insulin response below the threshold (as defined below) on two occasions, if their oral glucose-tolerance results were not completely normal,or both.

Relatives who tested positive for islet-cell antibodies and insulin antibodies and who had a first-phase insulin response above the threshold and normal glucose tolerance were defined as having intermediate risk (a five-year risk of 26 to 50 percent) and were deemed eligible for the ongoing oral insulin trial.

All randomized subjects were seen every six months, at which time an oral glucose-tolerance test was administered to assess glycemic status, the primary study end point. Mixed-meal tolerance tests were performed at base line, at years 1, 3, and 5, and at the end of the study. Intravenous glucose-tolerance testing was performed at years 2, 4, and 6 and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 3-45 years old who have an immediate family member with type 1 diabetes (such as a child, parent, or sibling)
* Individuals 3-20 years old who have an extended family member with type 1 diabetes (such as a cousin, niece, nephew, aunt, uncle, grandparent, or half-sibling)

Exclusion Criteria:

* To be eligible, a person must:
* Not have diabetes already.
* Have no previous history of being treated with insulin or oral diabetes medications.
* Have not received any prior therapy for prevention of type 1 diabetes such as insulin, nicotinamide, or immunosuppressive drugs (i.e. have not been involved in any previous clinical studies of these agents.)
* Have no known serious diseases.
* If you are a woman, you must not be planning to become pregnant during the course of the study. You will not be excluded from participation, but are not encouraged to volunteer in the first place if you plan to have a baby during the trial period).

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 711 (Actual)
Dates: Start 1994-02 (Actual); Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Rate of Type 1 Diabetes Per Year | Glucose tolerance is measured every 6 months for up to 6 years
  The rate of type 1 diabetes per year is calculated by dividing the number of participants who develop diabetes by the total number of years of follow-up. The diagnosis of diabetes is as defined by the American Diabetes Association (ADA) based on oral glucose testing or the presence of symptoms and unequivocal hyperglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Jay S. Skyler, MD, Study Chair — University of Miami
Locations (15):
- United States (14):
  - Childrens Hospital of Los Angeles, Division of Endocrinology, Los Angeles, California
  - University of California-San Francisco, Milberry Union East RM 405, 500 Parnassus Ave Box 0136, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Barbara Davis Center for Childhood Diabetes, Denver, Colorado
  - University of Florida Diabetes Research Center, Gainesville, Florida
  - DPT-1 Operations Coordinating Center, Miami, Florida
  - University of Miami School of Medicine, Jackson Medical Tower, Miami, Florida
  - Indiana University, James Whitcomb Riley Hospital for Children, 702 Barnhill Dr, Ste 5960, Indianapolis, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Naomi Berrie Diabetes Center, Columbia University, 1150 St. Nicholas Ave, New York, New York
  - Children's Hospital of Pittsburgh, Dept/Pediatric Endocrinology, 3705 5th Ave, Pittsburgh, Pennsylvania
  - University of Texas, Children's Medical Center, 6300 Harry Hines Ste 1200, Dallas, Texas
  - Virginia Mason Research Center, 1201 Ninth Avenue, Seattle, Washington
- Hospital for Sick Children, Division of Endocrinology, 555 University Ave, Rm 5110, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/dpt-1/?query=dpt-1
URL: https://repository.niddk.nih.gov/studies/dpt-1/?query=dpt-1

REFERENCES:
- [Background] Shah SC, Malone JI, Simpson NE. A randomized trial of intensive insulin therapy in newly diagnosed insulin-dependent diabetes mellitus. N Engl J Med. 1989 Mar 2;320(9):550-4. doi: 10.1056/NEJM198903023200902. PMID 2644534
- [Background] Keller RJ, Eisenbarth GS, Jackson RA. Insulin prophylaxis in individuals at high risk of type I diabetes. Lancet. 1993 Apr 10;341(8850):927-8. doi: 10.1016/0140-6736(93)91215-8. PMID 8096268
- [Background] Zhang ZJ, Davidson L, Eisenbarth G, Weiner HL. Suppression of diabetes in nonobese diabetic mice by oral administration of porcine insulin. Proc Natl Acad Sci U S A. 1991 Nov 15;88(22):10252-6. doi: 10.1073/pnas.88.22.10252. PMID 1946445
- [Result] Skyler JS, Krischer JP, Wolfsdorf J, Cowie C, Palmer JP, Greenbaum C, Cuthbertson D, Rafkin-Mervis LE, Chase HP, Leschek E. Effects of oral insulin in relatives of patients with type 1 diabetes: The Diabetes Prevention Trial--Type 1. Diabetes Care. 2005 May;28(5):1068-76. doi: 10.2337/diacare.28.5.1068. PMID 15855569
- [Result] Diabetes Prevention Trial--Type 1 Diabetes Study Group. Effects of insulin in relatives of patients with type 1 diabetes mellitus. N Engl J Med. 2002 May 30;346(22):1685-91. doi: 10.1056/NEJMoa012350. PMID 12037147
- [Derived] Barker JM, McFann KK, Orban T. Effect of oral insulin on insulin autoantibody levels in the Diabetes Prevention Trial Type 1 oral insulin study. Diabetologia. 2007 Aug;50(8):1603-6. doi: 10.1007/s00125-007-0694-0. Epub 2007 Jun 22. PMID 17583798
- [Derived] Johnson SB, Baughcum AE, Hood K, Rafkin-Mervis LE, Schatz DA; DPT-1 Study Group. Participant and parent experiences in the parenteral insulin arm of the diabetes prevention trial for type 1 diabetes. Diabetes Care. 2007 Sep;30(9):2193-8. doi: 10.2337/dc06-2422. Epub 2007 Jun 11. PMID 17563348
- See also: Website for the American Diabetes Association which also gives information about the DPT-1. — http://www.diabetes.org